CLINICAL TRIAL: NCT02097888
Title: Influence of Erythropoietin on Bone Marrow Microenvironment: A Pilot Study
Brief Title: Influence of Erythropoietin on Bone Marrow Microenvironment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kantonsspital Baselland Bruderholz (Other)
Responsible Party: Principal Investigator, PD Dr. med. Sandrine Meyer-Monard, PD Dr. med., Kantonsspital Baselland Bruderholz
Other Study IDs: KSBLB: 252/11
Record Dates: First submitted 2014-03-19; First posted 2014-03-27 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: Healthy Men and Non- Pregnant Women

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Samples Without DNA - samples retained, with no potential for DNA extraction from any retained samples (e.g., fixed tissue, plasma)
Oversight: Data Monitoring Committee: No

SUMMARY:
This will be a prospective observational study. The investigators will compare Erythropoietin (Epo) levels, erythropoiesis, and regulators of erythropoiesis, bone imaging and bone metabolism in healthy volunteers living at different altitudes.

ELIGIBILITY:
Inclusion Criteria:

* healthy men and non-pregnant women, ages ≥18-40 years and ≥ 60 years living in the predefined area
* Exclusion Criteria:
* Known bone pathology including osteoporosis, known haematological disease, known renal disease, heart insufficiency, pulmonal disease
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents living < 400m over sea level and >1500m over sea level
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2011-12; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Difference of EPO level between control groups | up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine Meyer-Monard, PD Dr. med., Principal Investigator — Kantonsspital Baselland / Bruderholz, Department of Medicine, Studienabteilung, CH-4101 Bruderholz
Locations (1):
- Kantonsspital Baselland / Bruderholz, Bruderholz, Switzerland